CLINICAL TRIAL: NCT06660602
Title: Perioperative Cerebral Function Assessment for Cardiac Surgery
Acronym: PEACE
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Shujuan Li, M.D., China National Center for Cardiovascular Diseases
Other Study IDs: 2024-2460
Record Dates: First submitted 2024-10-21; First posted 2024-10-28 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery
Keywords: cardiac surgery; stroke; cognitive function; delirium; risk factor; predictive model
MeSH Terms: conditions — Stroke; Delirium | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: cardiac surgery — All kinds of cardiac surgeries

SUMMARY:
Perioperative neurological complications in cardiovascular surgical procedures are associated with a significant risk of mortality and disability. This study is aimed at identifying the specific risk factors associated with these neurological complications during the perioperation and developing a comprehensive predictive model designed to enhance clinical decision-making and improve patient safety. The research is divided into three key phases: preoperative, intraoperative, and postoperative, each involving targeted evaluations and continuous monitoring to provide a thorough assessment of patient risk and outcomes.

DETAILED DESCRIPTION:
Before operation, a thorough assessment is conducted, encompassing a detailed analysis of participants' medical histories, demographic profiles, cerebrovascular structure, and cerebral function. These variables are systematically examined to identify risk factors for neurological complications.

Intraoperatively, real-time monitoring of cerebral blood flow and regional oxygen saturation is conducted using advanced techniques, including transcranial Doppler ultrasound and near-infrared spectroscopy, to evaluate the impact of surgical procedures on cerebral perfusion and oxygenation.

Postoperative monitoring emphasizes the identification of potential complications, such as cognitive dysfunction, seizures, delirium, and stroke. By integrating data from all stages during perioperation, the investigators want to develop a predictive model for perioperative brain function assessment. This model is intended to provide clinicians with a reliable tool for more precise risk assessment and timely intervention, thereby reducing the incidence of neurological complications and improving the prognosis for patients.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-80 years;
2. Patients undergoing cardiovascular surgical procedures;
3. Able to understand and comply with the clinical trial protocol requirements, and willing to sign the informed consent form.

Exclusion Criteria:

1. Inability to tolerate required diagnostic procedures, including neck CT angiography (CTA), head CT perfusion (CTP), or electroencephalography (EEG), due to underlying physical limitations or medical contraindications;
2. Severe renal insufficiency, characterized by a creatinine clearance of less than 30 mL/min (using the Cockcroft-Gault formula), serum creatinine levels exceeding twice the upper limit of normal, or any other form of clinically significant renal impairment;
3. Severe hepatic dysfunction, defined by ALT or AST levels greater than three times the upper limit of normal, or the presence of hepatic conditions such as acute or chronic hepatitis, cirrhosis, or other significant liver disorders;
4. Comorbid conditions that may compromise study participation or pose substantial risk to the patient, including, but not limited to, alcohol or substance abuse, malignancies, and severe diseases affecting the liver, kidneys, lungs, endocrine system (e.g., uncontrolled diabetes or thyroid disorders), or hematopoietic system;
5. Inability to cooperate with study procedures, whether due to cognitive, psychological, or physical factors that would impede compliance with protocol requirements;
6. Other conditions deemed unsuitable by the investigator, including any medical or non-medical factors that, in the investigator's assessment, may preclude safe or effective participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent cardiac surgeries
Sampling Method: Probability Sample
Enrollment: 1845 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Neurological complications within 7 (±3) days post-surgery including fatal or non-fatal stroke, coma, or movement disorders; cognitive dysfunction or delirium | From enrollment to the post-surgery within 7 (±3) days

CONTACTS AND LOCATIONS:
Overall Officials: Li Shujuan, MD, Study Director — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Department of Neurology, Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gerstenecker A, Norling AM, Jacob A, Lazar RM. Silent Brain Infarction, Delirium, and Cognition in Three Invasive Cardiovascular Procedures: a Systematic Review. Neuropsychol Rev. 2023 Jun;33(2):474-491. doi: 10.1007/s11065-022-09548-1. Epub 2022 Jul 8. PMID 35804216
- [Background] Sultan I, Bianco V, Kilic A, Jovin T, Jadhav A, Jankowitz B, Aranda-Michel E, D'angelo MP, Navid F, Wang Y, Thoma F, Gleason TG. Predictors and Outcomes of Ischemic Stroke After Cardiac Surgery. Ann Thorac Surg. 2020 Aug;110(2):448-456. doi: 10.1016/j.athoracsur.2020.02.025. Epub 2020 Mar 19. PMID 32199830
- [Background] Vermeer SE, Prins ND, den Heijer T, Hofman A, Koudstaal PJ, Breteler MM. Silent brain infarcts and the risk of dementia and cognitive decline. N Engl J Med. 2003 Mar 27;348(13):1215-22. doi: 10.1056/NEJMoa022066. PMID 12660385
- [Background] Gaudino M, Rahouma M, Di Mauro M, Yanagawa B, Abouarab A, Demetres M, Di Franco A, Arisha MJ, Ibrahim DA, Baudo M, Girardi LN, Fremes S. Early Versus Delayed Stroke After Cardiac Surgery: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2019 Jul 2;8(13):e012447. doi: 10.1161/JAHA.119.012447. Epub 2019 Jun 19. PMID 31215306
- [Background] Hillis LD, Smith PK, Anderson JL, Bittl JA, Bridges CR, Byrne JG, Cigarroa JE, Disesa VJ, Hiratzka LF, Hutter AM Jr, Jessen ME, Keeley EC, Lahey SJ, Lange RA, London MJ, Mack MJ, Patel MR, Puskas JD, Sabik JF, Selnes O, Shahian DM, Trost JC, Winniford MD. 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 Dec 6;124(23):e652-735. doi: 10.1161/CIR.0b013e31823c074e. Epub 2011 Nov 7. No abstract available. PMID 22064599